

REC Reference Number: 17/L0/0184 IRAS ID: 210709 Patient Identification Number for this trial: \_\_\_\_\_ **CONSENT FORM Title:** Distribution of cell-cell junction proteins in arrhythmic disorders. Name of Researcher: Angeliki Asimaki, PhD Cardiology Clinical Academic Group Cardiovascular and Genomics Research Institute City St. George's, University of London, Cranmer Terrace, London, SW17 ORE Please initial each box 1. I confirm that I have read and understand the information sheet dated version\_\_\_\_\_ or the above study and have had the opportunity to consider the information, ask questions and have these answered satisfactorily. 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. 3. I understand that relevant sections of any of my medical notes and data collected during the study may be looked at by responsible individuals from City St George's University of London, the NHS Trust or from regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records. 4. I understand that if the results from the smears I obtain using the at-home kit are different to the results of previous smears I provided at the hospital, my regular medical team may call me and arrange to bring my regular annual follow-up appointment forward. 5. I agree to take part in the above study. 6. I agree to a research team member or myself using a soft brush to obtain cells from the inside of my mouth 7. I agree to my anonymised data and/or results being used for future research 8. I agree to my samples being used as described in the information sheet 9. I agree to my GP being informed of my involvement [OPTIONAL]



| 10. I want to receive a copy of the results' summary once the study has been completed [OPTIONAL] | | |
|---|---|---|
| Name of Patient | Date | Signature |
| Name of person taking consent | <br>Date | <br>Signature |

When completed 1 for patient; 1 for researcher; 1 (original) to be kept with hospital notes